CLINICAL TRIAL: NCT07094828
Title: Integration of Augmented Visual Feedback Into Action Observation and Motor Imagery Therapy for Parkinson's Disease: A Randomized Controlled Trial
Brief Title: Integration of Augmented Visual Feedback in Action Observation and Motor Imagery Therapy for Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergamo (Other)
Collaborators: Fondazione Europea di Ricerca Biomedica Ferb Onlus (Other)
Responsible Party: Principal Investigator, Francesca Morganti, Associate Professor, University of Bergamo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0026841/25
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Action Observation; Motor Imagery; Technology; Physiotherapy; Gait Analysis
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researcher in charge of Data Analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation and Motor Imagery integrated with D-Wall technology (Experimental)
  Interventions: Other: AOMI with D-Wall
- Routine rehabilitative physiotherapy integrated with D-Wall technology (Active Comparator)
  Interventions: Other: Routine physiotherapy with D-Wall

INTERVENTIONS:
Other: AOMI with D-Wall — The intervention group will follow routine rehabilitative activity in the morning and will perform one hour of Action Observation and Motor Imagery training with augmented visual feedback (D-Wall) in the afternoon, three times a week.
  Each session will be conducted as follows: first AO (Action Observation), then MI (Motor Imagery). During the MI phase, participants will be asked to imagine the motor tasks and then perform them, receiving real-time augmented visual feedback provided by the digital mirror.
  Other Names: Action Observation and Motor Imagery integrated with D-Wall technology
  Arms: Action Observation and Motor Imagery integrated with D-Wall technology
Other: Routine physiotherapy with D-Wall — The control group will also follow routine rehabilitative activity in the morning, while in the afternoon they will perform motor training of the same duration, without Action Observation and Motor Imagery, but solely with augmented visual feedback (D-Wall), with the same weekly frequency.
  Other Names: Routine rehabilitative physiotherapy integrated with D-Wall technology
  Arms: Routine rehabilitative physiotherapy integrated with D-Wall technology

SUMMARY:
Improving movement control during rehabilitation is still a challenge for people with Parkinson's Disease, mainly because of the motor symptoms caused by the condition. However, new technologies offer promising ways to support therapy.

This clinical trial will test whether using TecnoBody® D-Wall technology integrated with two techniques (Action Observation and Motor Imagery) can improve physiotherapy outcomes for people with Parkinson's Disease.

The TecnoBody® D-Wall is a type of digital mirror that includes a 3D camera, pressure-sensitive platforms, and a screen. It shows a person's body movements in real time and gives visual feedback on joint mobility, balance, and how weight is distributed during movement.

Action Observation and Motor Imagery are two techniques already used in physiotherapy. Action Observation involves watching someone perform a movement, while Motor Imagery involves mentally rehearsing the movement before doing it. Studies have shown that both techniques activate the same brain areas involved in actual movement.

In this trial, after watching and imagining the movement, participants will perform the exercise in front of the D-Wall. This setup gives them real-time feedback to help improve how they move, a new approach for these techniques.

To see if this approach works, we will measure balance using a test validated for people with Parkinson's Disease and assess mobility using lab-based gait analysis, which tracks how a person walks.

Participants in the study will:

* Be receiving routine physiotherapy at a hospital that is specialized in Parkinson's Disease rehabilitation.
* Be randomly assigned to one of two groups: 1) One group will receive physiotherapy incorporating the D-Wall alongside Action Observation and Motor Imagery; 2) The other group will receive physiotherapy incorporating the D-Wall but, without Action Observation or Motor Imagery.
* Take part in therapy for up to four weeks, followed by another four weeks of monitoring, for a total of up to two months.
* Complete some initial tests to check if they are eligible for the study.

This study includes patients who have been diagnosed with idiopathic Parkinson's Disease and are undergoing rehabilitation as part of their usual hospital care. The intervention lasts as long as their regular hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic Parkinson's disease for at least 5 years;
* stable medication regimen for at least 4 weeks;
* no cognitive impairment according to the Mini-Mental State Examination;
* at stage ≤3 on the Hoehn & Yahr scale;
* provide informed consent to participate.

Exclusion Criteria:

* undergoing advanced therapies (e.g., deep brain stimulation or infusion pump therapy);
* unable to walk independently for at least 5 meters without assistive devices;
* substance abuse;
* with visual, orthopedic, or other medical conditions that could hinder the execution of activities;
* history of other neurological disorders (other than Parkinson's disease).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Dynamic postural control | at baseline, at the fourth week (end of the intervention period), and at the eighth week (follow-up).
  The Mini-Balance Evaluation Systems Test (Mini-BESTest) will be used to assess dynamic postural control.

SECONDARY OUTCOMES:
Moviment analysis | at baseline, at the fourth week (end of the intervention period), and at the eighth week (follow-up).
  Secondary outcomes will be obtained through instrumented motion analysis. Specifically, it will include spatiotemporal parameters and descriptive measures of the kinematics and dynamics of the hip, knee, and ankle joints.

IPD SHARING:
Plan to Share IPD: Undecided